CLINICAL TRIAL: NCT03015272
Title: Testing a Novel Speech Intervention in Minimally Verbal Children With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Gottfried Schlaug, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012P000344
Record Dates: First submitted 2016-01-29; First posted 2017-01-10 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Autism
Keywords: minimally-verbal; children; intervention; singing; music
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auditory-Motor Mapping Training (AMMT) (Experimental): Auditory-Motor Mapping Training (AMMT) is a novel, intonation-based intervention that is accompanied by simultaneous tapping each spoken syllable on tuned drums designed to help minimally verbal children between the ages of 5.5 and 12 years develop and/or improve speech output. AMMT is administered 1-on-1 for 45 min./day, 5 days/week (25 sessions) by researchers trained in this intervention.
  Interventions: Behavioral: Auditory-Motor Mapping Training
- Speech-Repetition Therapy (SRT) (Active Comparator): Speech-Repetition-Therapy (SRT) is a novel, non-intonation-based intervention designed to help minimally verbal children between the ages of 5.5 and 12 years develop and/or improve speech output. SRT is administered 1-on-1 for 45 min./day, 5 days/week (25 sessions) by researchers trained in this intervention. SRT serves as a control intervention to AMMT
  Interventions: Behavioral: Speech-Repetition Therapy

INTERVENTIONS:
Behavioral: Auditory-Motor Mapping Training — AMMT is a novel, intonation-based intervention that is accompanied by simultaneous tapping each spoken syllable on tuned drums, designed to help minimally verbal children between the ages of 5.5 and12.0 years develop and/or improve speech output. AMMT is administered 1-on-1 for 45 min./day, 5 days/week (25 sessions) by researchers trained in the method.
  Other Names: AMMT
  Arms: Auditory-Motor Mapping Training (AMMT)
Behavioral: Speech-Repetition Therapy — SRT is a novel, non-intonation-based intervention designed to help minimally verbal children between the ages of 5.5 and 12 years develop and/or improve speech output. SRT is administered 1-on-1 for 45 min./day, 5 days/week (25 sessions) by researchers trained in this intervention. SRT serves as a control intervention to AMMT.
  Other Names: SRT
  Arms: Speech-Repetition Therapy (SRT)

SUMMARY:
The goal of the Novel Language Intervention for minimally verbal children with Autism Spectrum Disorder (ASD) is to test the efficacy of one experimental treatment (AMMT) compared to baseline assessments and compare the AMMT efficacy to a control intervention (SRT), both treatments were designed to facilitate speech output in minimally verbal 5.5 to 12.0 year olds. This study aims to compare the two interventions (one intonation-based; the other non-intonation-based) in a single-blind, randomized controlled trial (RCT) that includes a comprehensive baseline assessment battery, 25 intensive 1-on-1 treatment sessions conducted 5 days/week, and a series of probe assessments administered at multiple timepoints pre-, during, and post-therapy.

Despite the complex needs of minimally verbal children with ASD and the wide variety of treatments available to address many of those needs, there is still a great need for effective methods that promote the development of speech sounds and facilitate the production of those sounds in this growing population. While the primary aim of this RCT is to investigate the effects of AMMTversus a control intervention (SRT) on minimally verbal children with ASD and compare the two interventions to determine whether one is more effective than the other, this study also aims to examine whether baseline cognitive skills, speech praxis, joint attention abilities and/or neural architecture can predict the effects of treatment with AMMT or SRT in minimally verbal children with ASD.

DETAILED DESCRIPTION:
The ability to communicate verbally is considered the most important prognostic indicator for children with ASD. If a child has not developed speech by age 5, it is generally considered unlikely that he or she will do so. Although a small number of cases of speech development in older children with ASD have been reported, the type and intensity of treatments used varied widely, suggesting little consensus regarding the likely mechanisms involved. A few preliminary studies have tested the efficacy of interventions that employed techniques such as orienting cues, behavioral strategies, and prompts for facilitating speech acquisition in minimally verbal children, though almost all tested their approaches in children under the age of 5 who would be classified as preverbal rather than minimally verbal.

Principal Investigator Gottfried Schlaug, MD, PhD oversees all aspects of study treatments for the interventional arm of this Autism Center of Excellence directed by Helen Tager-Flusberg of Boston University. The Intervention study's main objective is to compare the effectiveness of one novel treatment for minimally verbal children with autism spectrum disorders (ASD), Auditory-Motor Mapping Training (AMMT) to a control intervention termed Speech Repetition Therapy (SRT), both of which were developed and piloted in Dr. Schlaug's laboratory. The aim of the present study is to test whether one of those treatments is more effective than the other in a group of 5;5 to 12;0 year olds.

Participants will be screened and undergo several tests at Boston University's (BU) Autism Center of Excellence. Those found eligible for the intervention "Testing a novel speech intervention in minimally verbal children with ASD" will be enrolled and undergo testing at BU, participate in MRI scanning at Massachusetts General Hospital's (MGH) Martinos Imaging Center, and will then be randomly assigned to either the AMMT or SRT group for treatment at BIDMC. Before the intervention begins, participants will have up to 5 Baseline testing sessions (approx. 45-60 min./session) to (1) determine their ability to repeat a set of high-frequency 2-syllable words/phrases (e.g., Hello and All done), and (2) obtain an inventory of speech sounds that they are able to produce prior to treatment.

The intervention consists of 25 one-on-one therapy sessions during which children will be working toward producing (or approximating) a set of high-frequency 2-syllable words/phrases (e.g., "More, please", "Mommy", "All done", etc.). Progress will be monitored several times during the treatment phase as well as immediately after the 25 sessions and 4-weeks later. The total time commitment for the Intervention portion of the study will be approximately 6-8 weeks (i.e., approx. 1 week (±) for Baseline testing; approx. 5 weeks (5 sessions/week) for treatment; and approx. 1 week (±) for several mid- and post-treatment testing sessions). Upon completion of the intervention at BIDMC, participants will undergo post-treatment testing at BU and follow-up MRI at MGH's Martinos Imaging Center.

Results of this study will not only help determine if one of the two interventions is effective by comparing post-treatment assessments to baseline assessments but will also compare the experimental treatment (AMMT) versus the control treatment (SRT) to examine whether or not one is more effective than the other.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 5;6 and 12;0 years,
* have a diagnosis of ASD,
* be classified as "minimally verbal" (which is defined as having fewer than 20 spoken words/phrases used for functional communication),
* demonstrate minimal progress in speech acquisition despite having had at least 18 months of speech therapy,
* have no other significant neurological or psychiatric illnesses/disorders other than ASD
* have no major hearing impairment,
* have a nonverbal mental age over 18 months,
* be able to follow 1-step commands without prompting,
* be able to sit in a chair for more than 15 minutes at a time, and
* be able to imitate at least 2 speech sounds on command.
* Families must agree to:
* - attend testing and treatment sessions at BIDMC 5 days/week for approx. 6-8 weeks,
* - attend pre- and post-intervention testing at BU's Autism Center of Excellence,
* - pre- and post-intervention MRI scanning at MGH's Martinos Center, and
* - video-recording of testing and treatment sessions.
* - suspend all other extracurricular speech / language therapies for the duration of the study.

Exclusion Criteria:

* have a history of significant neurological or psychiatric disorder other than ASD that could interfere with this study as determined by PI;
* have a major hearing impairment,
* have a nonverbal mental age of less than 18 months,
* have undergone a significant amount of intonation-based therapy (more than 25 sessions) within the 12 months period prior to enrollment,
* are able to produce more 20 or more words used communicatively,
* are unable to imitate at least 2 speech sounds on command,
* cannot commit to pre- and post- intervention testing and MRI at BU and MGH,
* cannot commit to 11 weeks of testing and treatment at BIDMC,
* are not willing to be video-recorded.

Ages: 66 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2014-11; Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in approximately correct Consonant-Vowel Syllables between Best-Baseline and Post-25-session assessment | ≥3 Baseline Assessments (over 1 week) after randomization and before therapy initiation; 4 assessments during and after therapy period (after 10, 15, 20, 25 sessions), and one follow-up assessment 4 weeks after the End of Therapy (total period 11 weeks)
  Approximately correct consonant-vowel syllables of 30 target words/phrases (15 Trained; 15 Untrained) presented using visual clues during at least 3 baseline assessments, multiple interim assessments (after 10, 15, 20, 25 therapy sessions), and one post-treatment assessment (4 weeks after the end of therapy).

SECONDARY OUTCOMES:
Change in approximately correct Consonant-Vowel Syllables between Best-Baseline and Post-4-week follow-up assessment | ≥3 Baseline Assessments (over 1 week) after randomization and before therapy initiation; 4 assessments during and after therapy period (after 10, 15, 20, 25 sessions), and one follow-up assessment 4 weeks after the End of Therapy (total period 11 weeks)
  Approximately correct consonant-vowel syllables of 30 target words/phrases (15 Trained; 15 Untrained) presented using visual clues during at least 3 baseline assessments, multiple interim assessments (after 10, 15, 20, 25 therapy sessions), and one post-treatment assessment (4 weeks after the end of therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Schlaug, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center/Harvard Medical School
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston University, Autism Center of Excellence, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wan CY, Bazen L, Baars R, Libenson A, Zipse L, Zuk J, Norton A, Schlaug G. Auditory-motor mapping training as an intervention to facilitate speech output in non-verbal children with autism: a proof of concept study. PLoS One. 2011;6(9):e25505. doi: 10.1371/journal.pone.0025505. Epub 2011 Sep 29. PMID 21980480
- [Background] Wan CY, Schlaug G. Neural pathways for language in autism: the potential for music-based treatments. Future Neurol. 2010 Nov;5(6):797-805. doi: 10.2217/fnl.10.55. PMID 21197137
- [Background] Wan CY, Demaine K, Zipse L, Norton A, Schlaug G. From music making to speaking: engaging the mirror neuron system in autism. Brain Res Bull. 2010 May 31;82(3-4):161-8. doi: 10.1016/j.brainresbull.2010.04.010. Epub 2010 Apr 28. PMID 20433906
- [Background] Kasari C, Brady N, Lord C, Tager-Flusberg H. Assessing the minimally verbal school-aged child with autism spectrum disorder. Autism Res. 2013 Dec;6(6):479-93. doi: 10.1002/aur.1334. Epub 2013 Oct 29. PMID 24353165
- [Background] Tager-Flusberg H. Promoting communicative speech in minimally verbal children with autism spectrum disorder. J Am Acad Child Adolesc Psychiatry. 2014 Jun;53(6):612-3. doi: 10.1016/j.jaac.2014.04.005. No abstract available. PMID 24839879
- [Background] Chenausky K, Norton A, Tager-Flusberg H, Schlaug G. Auditory-Motor Mapping Training: Comparing the Effects of a Novel Speech Treatment to a Control Treatment for Minimally Verbal Children with Autism. PLoS One. 2016 Nov 9;11(11):e0164930. doi: 10.1371/journal.pone.0164930. eCollection 2016. PMID 27829034
- See also: Dr. Schlaug's lab website — http://www.musicianbrain.com
- See also: Boston University, Autism Center of Excellence — http://www.bu.edu/autism/current-research/autism-center-of-excellence/novel-language-intervention/